CLINICAL TRIAL: NCT07388199
Title: Effects of a Foot Core Training Program on Foot Pain, Function, and Pressure Pain Sensitivity in Patients With Fibromyalgia: A Quasi-Experimental Study.
Brief Title: Foot Core Intervention for Fibromyalgia
Acronym: FOOTCORE-FM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Collaborators: Universidad de León (Other)
Responsible Party: Principal Investigator, CARMEN GARCÍA GOMARIZ, principal investigator, University of Valencia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FOOTFIBRO_01
Record Dates: First submitted 2026-01-22; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Fibromyalgia; Foot Core
Keywords: Foot pain; Foot function; Pressure pain sensitivity; Quality of life
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Intervention Model Description: This study uses a single-group, pre-post quasi-experimental design, in which all participants receive the same intervention and outcomes are measured before and after the program. There is no control group or randomization.
Masking Description: This study uses partial masking. Participants were not blinded, as they were aware of their participation in an exercise-based intervention and the nature of the foot core training program. However, the outcome assessor was blinded to the study objectives and to the timing of the evaluations (baseline vs. post-intervention) to minimize assessment bias.
  The assessor responsible for collecting FHSQ scores and pressure pain threshold measurements did not have access to participant allocation information, intervention details, or previous results. This single-blind approach ensures that outcome measurements are performed objectively, reducing potential expectancy or observational bias typically associated with non-blinded participants in exercise studies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group Footcore (Experimental): The experimental group consisted of adults with medically diagnosed fibromyalgia who completed an eight-week supervised foot core training program (2 sessions/week, 45 minutes), including intrinsic foot strengthening and progressive balance tasks. All participants received the same intervention, with individualized load adjustment to ensure safety and prevent symptom exacerbation.
  Interventions: Other: Foot Core

INTERVENTIONS:
Other: Foot Core — Eight-week supervised foot core training (2×/week, 45 min) including mobility, intrinsic foot muscle strengthening, and progressive balance tasks. Exercises progressed from basic activation to standing and single-leg control. Load was individualized to prevent symptom exacerbation and ensure safe participation.

SUMMARY:
This quasi-experimental study was designed to evaluate the effects of an eight-week foot core training program on foot pain, foot function, and pressure pain sensitivity in individuals with fibromyalgia. Participants were recruited among individuals diagnosed with fibromyalgia according to the American College of Rheumatology (ACR) and the American Pain Society-American Academy of Pain Medicine (AAPT) criteria.

The intervention consisted of a structured foot core training program focused on strengthening the intrinsic foot musculature. Assessments were conducted before and after the intervention period. Outcome measures included foot pain and foot function assessed using the Foot Health Status Questionnaire (FHSQ), as well as pressure pain thresholds measured using mechanical algometry at six predefined rearfoot anatomical points.

DETAILED DESCRIPTION:
This quasi-experimental study was designed to evaluate the effects of an eight-week foot core training program on foot pain, foot function, and pressure pain sensitivity in individuals with fibromyalgia. Participants were recruited from individuals diagnosed with fibromyalgia in accordance with the criteria established by the American College of Rheumatology (ACR) and the American Pain Society-American Academy of Pain Medicine (AAPT).

The intervention consisted of a structured foot core training program aimed at strengthening the intrinsic musculature of the foot and was implemented over an eight-week period. The program was designed to be delivered in a systematic and progressive manner.

Assessments were performed prior to the initiation of the intervention and at the end of the eight-week training period. Outcome measures included foot pain and foot function, assessed using the Foot Health Status Questionnaire (FHSQ). Pressure pain sensitivity was evaluated using mechanical algometry, with pressure pain thresholds recorded at six predefined anatomical points of the rearfoot.

All measurements were conducted following standardized procedures and by trained personnel. The data collected were intended to examine changes in foot-related outcomes and pressure pain sensitivity following completion of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 65 years.
* Medical diagnosis of fibromyalgia according to the current American College of - Rheumatology (ACR) criteria and the AAPT criteria.
* Ability to understand instructions and complete all assessment procedures.
* Capacity to perform the exercise program without severe motor impairments that would limit participation.
* Voluntary agreement to participate and signed informed consent.

Exclusion Criteria:

* Severe comorbidities (e.g., cardiovascular, neurological, or systemic conditions) that could interfere with participation.
* Relevant pre-existing podiatric pathologies that may alter foot mechanics or confound outcomes.
* Pregnancy.
* Severe psychiatric disorders that could interfere with adherence or accurate outcome assessment.
* Inability to attend sessions or comply with study procedures.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2026-01-15 (Actual); Study Completion 2026-01-22 (Actual)

PRIMARY OUTCOMES:
Foot Pain (FHSQ Foot Pain Domain) | Baseline (Week 0) and Post-intervention (Week 8)
  Change in foot pain as measured by the Foot Health Status Questionnaire (Foot Pain domain).
  The Foot Health Status Questionnaire (FHSQ) is a validated, foot-specific patient-reported outcome measure. Scores range from 0 to 100, where higher scores indicate better foot health and less pain, and lower scores indicate worse foot pain. A score of 0 represents the worst possible foot pain, and a score of 100 represents no foot pain / best possible foot health.

SECONDARY OUTCOMES:
Pressure Pain Sensitivity (Pressure Pain Thresholds by Algometry) | Baseline (Week 0) and Post-intervention (Week 8)
  Change in pressure pain thresholds measured with a mechanical algometer (Fischer FDK/FDN).
  Pressure pain thresholds were assessed using a mechanical algometer (Fischer FDK/FDN). Pressure was applied gradually at a rate of 1 kg/s at six anatomical sites of the rearfoot (right and left sinus tarsi, medial malleolus, and lateral malleolus). Measurements were recorded in kilograms per square centimeter (kg/cm²). The measurement range was 0 to 11 kg/cm², where higher values indicate higher pressure pain thresholds and reduced mechanosensitivity, and lower values indicate greater pain sensitivity.
Vigor and General Health (FHSQ Domains) | Baseline (Week 0) and Post-intervention (Week 8)
  Change in vitality and general health as measured by the Foot Health Status Questionnaire (FHSQ).
  Vitality and general health were assessed using the corresponding domains of the Foot Health Status Questionnaire (FHSQ), a validated foot-specific patient-reported outcome measure. Each domain is scored on a scale ranging from 0 to 100, where higher scores indicate better vitality and better perceived general health, and lower scores indicate worse vitality and poorer perceived general health. A score of 0 represents the worst possible status, and a score of 100 represents the best possible status for each domain.
Physical Activity and Social Capacity (FHSQ Domains) | Baseline (Week 0) and Post-intervention (Week 8)
  Change in physical activity levels and social participation as measured by the Foot Health Status Questionnaire (FHSQ).
  Physical activity and social participation related to foot health were assessed using the corresponding domains of the Foot Health Status Questionnaire (FHSQ), a validated foot-specific patient-reported outcome measure. Each domain is scored on a scale ranging from 0 to 100, where higher scores indicate better physical activity levels and greater social participation, and lower scores indicate worse functional capacity. A score of 0 represents the worst possible status, and a score of 100 represents the best possible status for each domain.

CONTACTS AND LOCATIONS:
Overall Officials: Roi Painceira Villar, Phd, Principal Investigator — Universidad de León
Locations (1):
- Universitat de València, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sarzi-Puttini P, Giorgi V, Marotto D, Atzeni F. Fibromyalgia: an update on clinical characteristics, aetiopathogenesis and treatment. Nat Rev Rheumatol. 2020 Nov;16(11):645-660. doi: 10.1038/s41584-020-00506-w. Epub 2020 Oct 6. PMID 33024295
- [Background] Siracusa R, Paola RD, Cuzzocrea S, Impellizzeri D. Fibromyalgia: Pathogenesis, Mechanisms, Diagnosis and Treatment Options Update. Int J Mol Sci. 2021 Apr 9;22(8):3891. doi: 10.3390/ijms22083891. PMID 33918736
- [Background] Hoegh M. Pain Science in Practice (Part 3): Peripheral Sensitization. J Orthop Sports Phys Ther. 2022 Jun;52(6):303-306. doi: 10.2519/jospt.2022.11202. PMID 35647877
- [Background] Smith SB, Maixner DW, Fillingim RB, Slade G, Gracely RH, Ambrose K, Zaykin DV, Hyde C, John S, Tan K, Maixner W, Diatchenko L. Large candidate gene association study reveals genetic risk factors and therapeutic targets for fibromyalgia. Arthritis Rheum. 2012 Feb;64(2):584-93. doi: 10.1002/art.33338. PMID 21905019
- [Background] Beiner E, Lucas V, Reichert J, Buhai DV, Jesinghaus M, Vock S, Drusko A, Baumeister D, Eich W, Friederich HC, Tesarz J. Stress biomarkers in individuals with fibromyalgia syndrome: a systematic review with meta-analysis. Pain. 2023 Jul 1;164(7):1416-1427. doi: 10.1097/j.pain.0000000000002857. Epub 2023 Jan 5. PMID 36728497
- [Background] Sun N, Hartmann R, Lecher J, Stoldt M, Funke SA, Gremer L, Ludwig HH, Demuth HU, Kleinschmidt M, Willbold D. Structural analysis of the pyroglutamate-modified isoform of the Alzheimer's disease-related amyloid-beta using NMR spectroscopy. J Pept Sci. 2012 Nov;18(11):691-5. doi: 10.1002/psc.2456. Epub 2012 Sep 24. PMID 23001756
- [Background] Bennett PJ, Patterson C, Wearing S, Baglioni T. Development and validation of a questionnaire designed to measure foot-health status. J Am Podiatr Med Assoc. 1998 Sep;88(9):419-28. doi: 10.7547/87507315-88-9-419. PMID 9770933